CLINICAL TRIAL: NCT05931627
Title: The Implications of Tourniquet Use on Early Quadriceps Function in Anterior Cruciate Ligament Reconstructions: A Randomized Controlled Trial
Brief Title: Tourniquet Use in Anterior Cruciate Ligament Repair
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SPORT177
Record Dates: First submitted 2023-05-31; First posted 2023-07-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: ACL - Anterior Cruciate Ligament Deficiency; ACL Injury; ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: Treating physicians and subjects will be blinded to treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Patients undergoing patellar bone-tendon-bone autograft ACL reconstruction with a tourniquet used for the duration of the case.
- Treatment/Intervention (Active Comparator): Patients undergoing ACL reconstruction with a tourniquet used only during patellar bone-tendon-bone autograft harvest, for a maximum of 20 minutes.
  Interventions: Procedure: Patients undergoing ACL reconstruction with or without a tourniquet

INTERVENTIONS:
Procedure: Patients undergoing ACL reconstruction with or without a tourniquet — Patients undergoing ACL reconstruction with or without a tourniquet
  Arms: Treatment/Intervention

SUMMARY:
The purpose of this study is to assess the intra-operative and post-operative effects of tourniquet use during ACL reconstruction. We hypothesize that:

1. Limited tourniquet use will not significantly impact arthroscopic visualization nor the time it takes to complete an ACL reconstruction.
2. Limited tourniquet use will lead to significantly less patient pain intra-operatively and in the immediate peri-operative period.
3. Patients who undergo an ACL reconstruction with limited tourniquet use will have earlier return of quadriceps functions as compared to those undergoing reconstruction with the use of a tourniquet.

DETAILED DESCRIPTION:
Type of Study Double-blinded randomized controlled clinical trial

Group 1 (Control): Patients undergoing patellar bone-tendon-bone autograft ACL reconstruction with a tourniquet used for the duration of the case.

Group 2 (Treatment/Intervention, if applicable): Patients undergoing ACL reconstruction with a tourniquet used only during patellar bone-tendon-bone autograft harvest, for a maximum of 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing an arthroscopic assisted ACLR using a bone-tendon-bone patellar tendon autograft.
2. 18 years or older
3. English speaking

Exclusion Criteria:

1. Concomitant procedures (e.g., osteotomy or other ligamentous reconstructions) other than chondroplasty, partial meniscectomy or meniscal repair
2. Medical contraindications to epinephrine or TXA use.
3. Hemophilia or other predisposition for bleeding
4. Does not follow study protocol in regard to regional anesthesia, TXA, epinephrine use in the arthroscopy fluid and post-operative rehabilitation.
5. Participation in physical therapy at any facility other than the OrthoCarolina Randolph, Matthews or South Park locations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Limb symmetry index (LSI) | 6 months
  Limb symmetry index (LSI) of the peak torque of the quadriceps

SECONDARY OUTCOMES:
Arthroscopic visibility | during surgery
  Arthroscopic visibility
Operative time | during surgery
  Operative time
Intra-operative opioid requirements | during surgery
  Intra-operative opioid requirements (in morphine milligram equivalents (MMEs)
PACU opioid requirements | during surgery
  PACU opioid requirements (MMEs)
Post-operative pain in PACU | during surgery
  Post-operative pain in PACU measured by a Numeric Rating Scale
LSI of peak strength and rate of torque development of the quadriceps | 6 weeks
  LSI of peak strength and rate of torque development of the quadriceps at 6 weeks, 3 months and 6 months as measured using a Tindeq Progressor 3000 dynamometer
LSI of peak strength and rate of torque development of the quadriceps | 6 months
  LSI of peak strength and rate of torque development of the quadriceps at 6 weeks, 3 months and 6 months as measured using a Tindeq Progressor 3000 dynamometer
Quadriceps circumference | preoperative, 2 weeks, 6 weeks, 3 months and 6 months
  Quadriceps circumference (at the proximal pole of the patella with the knee in extension) at 2 weeks, 6 weeks, 3 months and 6 months post-operatively, as compared to pre-operatively.
Number of days post-operatively until the patient can complete a straight leg raise with no extensor lag at physical therapy. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Number of days post-operatively until the patient can complete a straight leg raise with no extensor lag at physical therapy.
Number of days post-operatively until the patient can actively hyper-extend their knee at physical therapy. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Number of days post-operatively until the patient can actively hyper-extend their knee at physical therapy.
IKDC and the Marx Activity Rating Scale scores | 6 weeks
  subjective knee evaluation
IKDC and the Marx Activity Rating Scale scores | 1 year
  subjective knee evaluation
Limb symmetry index (LSI) | 6 weeks
  Limb symmetry index (LSI) of the peak torque of the quadriceps
Limb symmetry index (LSI) | 3 months
  Limb symmetry index (LSI) of the peak torque of the quadriceps

OTHER OUTCOMES:
Sex | preoperative
  Sex
Race | preoperative
  Race
Ethnicity | preoperative
  Ethnicity
Body Mass Index (BMI) | preoperative
  Body Mass Index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Riboh, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina Research Institute, Inc., Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grassi A, Carulli C, Innocenti M, Mosca M, Zaffagnini S, Bait C; SIGASCOT Arthroscopy Committee. New Trends in Anterior Cruciate Ligament Reconstruction: A Systematic Review of National Surveys of the Last 5 Years. Joints. 2018 Sep 27;6(3):177-187. doi: 10.1055/s-0038-1672157. eCollection 2018 Sep. PMID 30582107
- [Background] Hooper J, Rosaeg OP, Krepski B, Johnson DH. Tourniquet inflation during arthroscopic knee ligament surgery does not increase postoperative pain. Can J Anaesth. 1999 Oct;46(10):925-9. doi: 10.1007/BF03013125. PMID 10522577
- [Background] Reda W, ElGuindy AMF, Zahry G, Faggal MS, Karim MA. Anterior cruciate ligament reconstruction; is a tourniquet necessary? A randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2016 Sep;24(9):2948-2952. doi: 10.1007/s00167-015-3582-z. Epub 2015 Mar 19. PMID 25786826
- [Background] Kuo LT, Yu PA, Chen CL, Hsu WH, Chi CC. Tourniquet use in arthroscopic anterior cruciate ligament reconstruction: a systematic review and meta-analysis of randomised controlled trials. BMC Musculoskelet Disord. 2017 Aug 22;18(1):358. doi: 10.1186/s12891-017-1722-y. PMID 28830402
- [Background] Struijk-Mulder MC, Ettema HB, Verheyen CC, Buller HR. Deep vein thrombosis after arthroscopic anterior cruciate ligament reconstruction: a prospective cohort study of 100 patients. Arthroscopy. 2013 Jul;29(7):1211-6. doi: 10.1016/j.arthro.2013.04.015. PMID 23809456
- [Background] Janssen RP, Reijman M, Janssen DM, van Mourik JB. Arterial complications, venous thromboembolism and deep venous thrombosis prophylaxis after anterior cruciate ligament reconstruction: A systematic review. World J Orthop. 2016 Sep 18;7(9):604-17. doi: 10.5312/wjo.v7.i9.604. eCollection 2016 Sep 18. PMID 27672574
- [Background] Mingo-Robinet J, Castaneda-Cabrero C, Alvarez V, Leon Alonso-Cortes JM, Monge-Casares E. Tourniquet-related iatrogenic femoral nerve palsy after knee surgery: case report and review of the literature. Case Rep Orthop. 2013;2013:368290. doi: 10.1155/2013/368290. Epub 2013 Nov 26. PMID 24371536
- [Background] Lee YG, Park W, Kim SH, Yun SP, Jeong H, Kim HJ, Yang DH. A case of rhabdomyolysis associated with use of a pneumatic tourniquet during arthroscopic knee surgery. Korean J Intern Med. 2010 Mar;25(1):105-9. doi: 10.3904/kjim.2010.25.1.105. Epub 2010 Feb 26. PMID 20195412
- [Background] Nicholas SJ, Tyler TF, McHugh MP, Gleim GW. The effect on leg strength of tourniquet use during anterior cruciate ligament reconstruction: A prospective randomized study. Arthroscopy. 2001 Jul;17(6):603-7. doi: 10.1053/jars.2001.24854. PMID 11447547
- [Background] Arciero RA, Scoville CR, Hayda RA, Snyder RJ. The effect of tourniquet use in anterior cruciate ligament reconstruction. A prospective, randomized study. Am J Sports Med. 1996 Nov-Dec;24(6):758-64. doi: 10.1177/036354659602400610. PMID 8947397
- [Background] Merry K, Napier C, Chung V, Hannigan BC, MacPherson M, Menon C, Scott A. The Validity and Reliability of Two Commercially Available Load Sensors for Clinical Strength Assessment. Sensors (Basel). 2021 Dec 16;21(24):8399. doi: 10.3390/s21248399. PMID 34960492
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686